CLINICAL TRIAL: NCT02855879
Title: Evaluation of the Prevalence of anomalIes of Glucose Metabolism in Patients Undergoing a Coronary Artery Bypass Graft, Consequences for Morbi/Mortality in the Short and Medium Term
Brief Title: Evaluation of the Prevalence of anomalIes of Glucose Metabolism in Patients Undergoing a Coronary Artery Bypass Graft (CABG)
Acronym: IMPACT
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: VERGES 2014
Record Dates: First submitted 2016-07-28; First posted 2016-08-04 (Estimated); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Anomalies in Glucose Metabolism; Coronary Artery Bypass Graft

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- CAD patients
  Interventions: Other: Collection of biological data; Other: Collection of clinical data

INTERVENTIONS:
Other: Collection of biological data
Other: Collection of clinical data

SUMMARY:
The aim of this study is to determine the prevalence of diabetes and non-diabetic glucose metabolism anomalies (glucose intolerance, non-diabetic fasting hyperglycaemia in patients about to undergo coronary artery bypass grafting (CABG).

In addition, the effect of these anomalies on post CABG morbi/mortality in the short term will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* persons who have provided oral consent
* patients about to undergo coronary artery bypass grafting
* age >18 years

Exclusion Criteria:

* persons without national health insurance cover
* Adults under guardianship
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients about to undergo coronary artery bypass grafting
Sampling Method: Non-Probability Sample
Enrollment: 286 (Actual)
Dates: Start 2015-04-08 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-06-05 (Actual)

PRIMARY OUTCOMES:
Percentage of glucose anomalies (non-diabetic fasting hyperglycaemia, glucose intolerance, diabetes) in CAD patients about to undergo coronary artery bypass grafting. | Change from inclusion to week 2 and up to month 3

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France